CLINICAL TRIAL: NCT07135505
Title: The Effect of Early Time-Restricted Eating on Cardiometabolic Health and Circadian Rhythms in Hypertensive Older Adults With Habitual Prolonged Eating Window
Brief Title: Early Time-Restricted Eating in Older Adults With Hypertension
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: UAB Nutrition Obesity Research Center (Unknown)
Responsible Party: Principal Investigator, Yi Lin, Instructor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-300013053; UAB NORC Pilot Grant (Other Grant/Funding Number: UAB Nutrition Obesity Research Center Pilot/Feasibility Grant Program)
Record Dates: First submitted 2025-08-14; First posted 2025-08-22 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-12

CONDITIONS: Hypertension; Eating Behaviors
MeSH Terms: conditions — Hypertension; Feeding Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Early time-restricted eating
  Interventions: Behavioral: Early time-restricted eating
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Early time-restricted eating — The participants will be asked to fast for a target of 16 hours per day (eat ad libitum within the 8-hour eating window, starting between 6:30-8:30 am), 6 days/week for 12 weeks. Participants will be allowed to consume calorie-free beverages, sugar-free gum, and will be encouraged to drink plenty of water throughout the entire intervention period.
  Arms: Intervention

SUMMARY:
The purpose of this study is to find out how early time-restricted eating affects body rhythms and improves cardiometabolic health in older adults.

ELIGIBILITY:
Inclusion Criteria:

* Consent to participate in the study
* Men and women ≥ 60 years old
* Average office systolic BP ≥130 mmHg
* Self-reported ≥12 hours eating period per day of at least 5 days/week
* Stable health history over the past 2 months

Exclusion Criteria:

* Fasting >12 hours per day
* Actively trying to lose weight by participating in formal weight loss program or significantly restricting calorie intake
* Have lost ≥ 10 pounds in last 3 months
* Unable to wake up at a regular time between 6-8 am
* Perform overnight shift work more than 1day/week on average
* Resting heart rate of >120 beats per minute, systolic blood pressure > 180 mmHg and/or diastolic blood pressure of > 100 mmHg
* Have been diagnosed with diabetes
* On insulin or diabetes medication
* Unstable angina, heart attack or stroke in the past 3 months
* Continuous use of supplemental oxygen to manage a chronic pulmonary condition or heart failure
* Pregnant or breastfeeding
* Rheumatoid arthritis, Parkinson's disease or currently on dialysis
* Current diagnosis of a major psychiatric condition that would impair study participation
* Severe gastrointestinal disease, major gastrointestinal surgery, or active gallstone disease
* Active treatment for cancer in the past year
* Taking medications that preclude fasting for 16 hours (e.g. must be taken with food at least 12 hours apart)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood glucose | Baseline and 12 weeks
  measured by the continuous glucose monitor
Heart rate variability | Baseline and 12 weeks
  measured by the Holter monitor
Systolic Blood pressure | Baseline and 12 weeks
  measured by the ambulatory blood pressure monitor

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided
IPD may not be shared due to concerns regarding participant privacy and the sensitive nature of the health-related data collected.